CLINICAL TRIAL: NCT03712189
Title: The Utility of LifeFlow Rapid Fluid Infuser in Critical and Non-critical Pediatric Patients: a Mixed-method Pilot Study Protocol
Brief Title: LifeFlow Fluid Study- Non- Critical Pediatric Patients Having a Trans Abdominal Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: 410 Medical (Industry); Atlanta Pediatric Device Consortium (Other)
Responsible Party: Principal Investigator, Todd P Chang, MD MAcM, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHLA-18-00188
Record Dates: First submitted 2018-10-11; First posted 2018-10-19 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Dehydration in Children; Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Alaris Pump (No Intervention): Participants will receive IV fluids delivered by the Alaris IV Pump (standard of care) until their bladder is full.
- LifeFlow (Experimental): Participants will receive IV fluids delivered by the LifeFlow Fluid Device until their bladder is full.
  Interventions: Device: LifeFlow

INTERVENTIONS:
Device: LifeFlow — The LifeFlow® is a hand-operated rapid infuser designed to administer fluids to patients by a single user, for clinical situations in which a large volume or rapid infusion of fluid or colloid is required. The device delivers fluid in 10mL increments with each complete handle compression, which refills during release, automating a push-pull mechanism. The syringe then automatically refills with handle release.
  Arms: LifeFlow

SUMMARY:
This is an unblinded, randomized control study examining two fluid delivery modalities for non-critical female patients with a planned transabdominal pelvic ultrasound requiring intravenous fluid boluses.

DETAILED DESCRIPTION:
Subjects be identified during their clinical course in the ED and will be randomized to either the LifeFlow® fluid delivery or an IV fluid bolus through the Alaris® pump (standard of care). IV fluids will be provided until the subject notes the sensation of a full bladder, at which point, the standard of care clinical practice is to perform the ultrasound. The transabdominal pelvic ultrasound requires a full bladder for optimal visualization of the ovaries, adnexa, and uterus, and is the only alternative to a transvaginal pelvic ultrasound for virginal young women. All other clinical care is per standard of care. The only research component is the randomization and data collection.

ELIGIBILITY:
Inclusion Criteria:

* Female patients older than 1 month and less than 18 years
* Patients require IV crystalloid bolus fluids before a pelvic ultrasound

Exclusion Criteria:

* Known cardiac insufficiency or significant cardiac surgery
* Hepatic insufficiency
* Renal insufficiency
* Any known fluid overload states (ascites, pulmonary edema)
* On any diuretic or antihypertensive therapy
* Known pregnancy

Ages: 1 Month to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd P Chang, MD, Principal Investigator — Children's Hospital Los Angeles; Ara Festekjian, MD, Study Director — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kline M, Crispino L, Bhatnagar A, Panchal RA, Auerbach M. A Randomized Single-Blinded Simulation-Based Trial of a Novel Method for Fluid Administration to a Septic Infant. Pediatr Emerg Care. 2021 Jun 1;37(6):e313-e318. doi: 10.1097/PEC.0000000000001583. PMID 30106868

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alaris Pump | LifeFlow
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alaris Pump | LifeFlow | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.6 (2.9) | 13.9 (3.5) | 13.8 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Duration- Ultrasound Ordered to Completed
Description: The primary outcome variable is the duration (minutes) of time from when the ultrasound was ordered to the completion time of the ultrasound.
Time Frame: From ED (Emergency Department) arrival to discharge/admission, less than 12 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Alaris Pump | LifeFlow
Number analyzed (Participants) | 15 | 15
minutes | 154.4 (53.2) | 114.8 (31.9)

2. Secondary Outcome: Total IV Fluid (mL)
Description: Total IV fluid administered before ultrasound
Time Frame: From ED arrival to discharge/admission, less than 12 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Alaris Pump | LifeFlow
Number analyzed (Participants) | 15 | 15
mL | 1612.9 (654.4) | 1482.7 (676.3)

3. Secondary Outcome: Duration- Full Bladder
Description: Fluid initiation and subjective sensation of full bladder
Time Frame: From ED arrival to discharge/admission, less than 12 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Alaris Pump | LifeFlow
Number analyzed (Participants) | 15 | 15
minutes | 61.9 (43.6) | 26.9 (18.9)

ADVERSE EVENTS:
Time Frame: 6 months
Description: All subjects are not at risk of death (as part of inclusion criteria)
Arm/Group | Alaris Pump | LifeFlow
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT03712189/Prot_SAP_000.pdf